CLINICAL TRIAL: NCT04309591
Title: Cytosorb Therapy in Cardiac Surgery - a Retrospective Study of Hemoadsorption in Patients With Endocarditis
Brief Title: Cytosorb Therapy in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01740; ch19Santer
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Cardiopulmonary Surgery; Endocarditis; Peri-operative Cytokines Levels
Keywords: cytokine clearance; cardiac surgery; CytoSorb; cytokine removal
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CytoSorb haemoadsorption (HA) device — CytoSorb® cartridges contain biocompatible sorbent polystyrene divinylbenzene beads coated with polyvinylpyrrolidone, capable of removing inflammatory molecules (eg Interleukin). The cartridge is inserted in a cardio-pulmonary bypass circuit to remove inflammatory molecules during cardiac surgery .

SUMMARY:
Cardiopulmonary surgery is associated with inflammatory responses that can lead to systemic inflammatory responses (SIRS), organ dysfunction (MOD) and death especially in patients with endocarditis. Cytokine removal might therefore improve outcomes of patients undergoing cardiac surgery. CytoSorb is a device designed to remove cytokine (IL-6, IL-10, TNFalpha) from the blood to reduce immune reactions. This trial investigates the use of CytoSorb during cardiac surgery in patients with endocarditis at the University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

* patients with endocarditis undergoing cardiac surgery with cardio-pulmonary bypass circuit

Exclusion Criteria:

* denial of consent for data use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with endocarditis undergoing cardiac surgery with cardio-pulmonary bypass circuit at the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
In-Hospital mortality | during hospital stay for cardiac surgery from admission until discharge (approximately 15 days)
  In-Hospital mortality (number of deaths) of patients with endocarditis undergoing cardiac surgery and intra-operative CytoSorb haemoadsorption

SECONDARY OUTCOMES:
time in intensive care unit (days) | during hospital stay for cardiac surgery from admission until discharge (approximately 15 days)
  time in intensive care unit (days)
In-Hospital time (days) | hospital stay for cardiac surgery from admission until discharge (approximately 15 days)
  In-Hospital time (days)

CONTACTS AND LOCATIONS:
Overall Officials: David Santer, Dr. med, Principal Investigator — Universitätsspital Basel, Herzchirurgie
Locations (1):
- Klinik für Herzchirurgie, Universitätsspital Basel, Basel, Switzerland